CLINICAL TRIAL: NCT05762757
Title: Patient-centered Educational Material to Improve Colposcopy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Association of Obstetricians and Gynecologists (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202208064
Record Dates: First submitted 2023-02-20; First posted 2023-03-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cervical Cancer Screening
Keywords: cervical cancer screening; colposcopy; patient education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colposcopy educational material (Experimental): Participants will complete a 9-question quiz that will assess knowledge of colposcopy. They will then view the colposcopy educational material and answer the same 9-question quiz to assess their knowledge of colposcopy. Participants will complete the Acceptability Intervention Measure, the Intervention Appropriateness Measure, and the Feasibility of Intervention Measure. Participants will also be asked whether the educational material influences their intention to adhere to colposcopy.
  Interventions: Other: Colposcopy educational material

INTERVENTIONS:
Other: Colposcopy educational material — -Will consist of a handout featuring education and information regarding colposcopies.

SUMMARY:
The long-term goal is to develop, test, and disseminate a social needs navigator intervention that improves colposcopy adherence. Based on stakeholder feedback, this study addresses the need to include patient-centered educational material to the navigator program in order to improve patients' health literacy regarding cervical cancer prevention.

DETAILED DESCRIPTION:
The investigators will evaluate the effectiveness of the colposcopy educational material. The investigators aim to recruit 25 newly referred colposcopy patients before their appointment, ask them to take a 5-minute test about their knowledge of colposcopy, have them view an online demo of the educational resources, and then retake the test.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Abnormal cervical screen confirmed by cytology or pathology
* Referred to Washington University School of Medicine (WUSM) colposcopy clinic

Exclusion Criteria:

* History of cervical cancer
* Unable to consent

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Change in participant knowledge of colposcopy | Prior to viewing educational material and after viewing educational material (Day 1)
  -9 question questionnaire that will assess patient knowledge of colposcopy

SECONDARY OUTCOMES:
Acceptability of educational material as measured by the Acceptability of Intervention Measure | Day 1
  This is a 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely disagree-completely agree). Mean score is calculated.
Appropriateness of educational material as measured by the Intervention Appropriateness Measure | Day 1
  This is a 4-item measure of perceived intervention appropriateness. Items are measured on a 5-point Likert scale (Completely disagree-completely agree). Mean score is calculated.
Feasibility of educational material as measured by the Feasibility of Intervention Measure | Day 1
Number of participants who stated that the educational material will influence their intention to adhere to colposcopy | Day 1
  This is a 4-item measure of perceived intervention feasibility. Items are measured on a 5-point Likert scale (Completely disagree-completely agree). Mean score is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Kuroki, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu